CLINICAL TRIAL: NCT00634816
Title: Cross-sectional Study of Bone Mineral Density in Adult Survivors of Solid Pediatric Cancers
Brief Title: Bone Mineral Density in Adult Survivors of Solid Pediatric Cancers
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Timothy Damron, M.D., Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: Cross Sectional
Record Dates: First submitted 2008-03-04; First posted 2008-03-13 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Regional Osteoporosis as a Result of Chemotherapy
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chemotherapy recipients: Subjects who have undergone chemotherapy will receive DXA scan
  Interventions: Radiation: DXA Scan

INTERVENTIONS:
Radiation: DXA Scan — The patients will undergo total body, spine, proximal femoral, and forearm DEXA testing in a standardized fashion. Patients who have undergone limb surgery or irradiation to an extremity for local disease control will also undergo selected site DEXA or pQCT scanning, depending upon the site, of the affected extremity and the identical site on the contra-lateral extremity.

SUMMARY:
Specific subgroups of children who survive treatment for childhood malignancies have been shown to develop relative osteopenia following chemotherapy and are felt to be at risk for developing osteoporosis later in life due to their inability to reach peak bone mass during childhood.

DETAILED DESCRIPTION:
Specific subgroups of children who survive treatment for childhood malignancies have been shown to develop relative osteopenia following chemotherapy and are felt to be at risk for developing osteoporosis later in life due to their inability to reach peak bone mass during childhood. However, currently, there is no conclusive evidence that survivors of pediatric solid malignancies are at risk for these problems due to small numbers of patients analyzed. Our SUNY Upstate Medical University Pediatric Oncology Long-term Follow-up Clinic has recently established a coalition of other upstate New York cancer centers which allows access to a large number of these patients. The purpose is to perform a cross-sectional study of bone mineral density using dual-energy X-ray absorptiometry (DEXA) in adult survivors of solid pediatric tumors. The primary hypothesis is that pediatric solid cancer survivors will demonstrate significantly lower bone mineral density (BMD) compared to established age group controls. Identification of these patients as high risk for development of osteoporosis will allow clinical trials using novel and established agents.

This study has been ongoing for 5 years. To date there have been no problems with the conduct of this study. A total of 38 subjects that have been enrolled. Analysis of research to date reveals that solid tumor survivors are at increased risk for early osteopenia/osteoporosis. No subjects have withdrawn or been excluded for any reason other than inclusion/exclusion criteria since inception of the study. The study will be ongoing for recruitment of subjects and analysis.

There was one amendment made to the protocol. The amendment was to increase the upper age of the subjects to 40 years. This amendment was made due to that although our multivariate analysis showed a relationship with number of chemotherapy drugs, our statistical power to examine according to multiple other variables, such as individual diagnosis, was limited by the relatively small numbers of patients.

An article was submitted to the Journal of Pediatric Hematology Oncology and printed in the May 2005 issue.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the SUNY Upstate Medical Center Pediatric Oncology Long-term Survivor Clinic who were treated for solid tumors and lymphomas with chemotherapy beginning at age less than 16 will be recruited for participation. Patients must be less than 40 years of age to participate.

Exclusion Criteria:

* Patients treated for Acute Lymphocytic Leukemia (ALL) and those who received cranial irradiation or total body irradiation (groups already known to be at high risk for osteoporosis) will be excluded. In addition, any patient who received non-autologous bone marrow transplant will be excluded, as these patients may have graft versus host disease (also known to be associated with osteopenia).

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be recruited from the Oncology Clinic by one of the sub-investigators.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2003-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Osteoporosis after chemotherapy | April 2003-April 2006
  Does chemotherapy increase the risk of osteoporosis in patients

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Damron, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States